CLINICAL TRIAL: NCT04464200
Title: A Phase I Study of CD19-Targeted 19(T2)28z1xx Chimeric Antigen Receptor (CAR) Modified T Cells in Adult Patients With Relapsed or Refractory B-cell Malignancies
Brief Title: 19(T2)28z1xx Chimeric Antigen Receptor (CAR) T Cells in People With B-Cell Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-167
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Transformed Follicular Lymphoma to Diffuse Large B Cell Lymphoma; Chronic Lymphocytic Leukemia; Indolent Non-Hodgkin Lymphoma; Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia; Burkitt's Lymphoma; Primary CNS Lymphoma
Keywords: 19(T2)28z1XX CAR T cells; 20-167
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Burkitt Lymphoma

STUDY DESIGN:
Intervention Model Description: This is a standard phase I open-label dose-escalation trial. Cohorts of 3-6 patients will be infused with escalating doses of 19(T2)28z1XX CAR T cells to establish the MTD. There are 4 planned dose levels with one additional de-escalation dose level. A 3+3 design will be used to establish the RP2D. Once the RP2D is determined, the study will open to Dose Expansion phase and up to 12 patients with B-cell non-Hodgkin lymphoma (same eligibility criteria as the dose-escalation phase).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 19(T2)28z1xx CAR T cells (Experimental): Cohorts of 3-6 patients will be infused with escalating doses of 19(T2)28z1XX CAR T cells to establish the RP2D. There are 4 planned flat-dose levels: 25x10^6, 50 x 10^6, 100 x 10^6 and 200 x 10^6 CAR T cells and one de-escalation dose: 12.5 x 10^6 CAR T cells. A standard 3+3 dose escalation design will be implemented starting from dose 1.
  Interventions: Drug: 19(T2)28z1xx CAR T cells

INTERVENTIONS:
Drug: 19(T2)28z1xx CAR T cells — 2-7 days following the completion of the conditioning chemotherapy, patients will receive the CAR- T cells by IV infusion over 1-3 days depending on the dose level and formulation of the final CAR- T cells.

SUMMARY:
The purpose of this study is to test the safety of 19(T2)28z1xx CAR T cells in people with relapsed/refractory B-cell cancers. The researchers will try to find the highest dose of 19(T2)28z1xx CAR T cells that causes few or mild side effects in participants. Once they find this dose, they can test it in future participants to see if it is effective in treating their relapsed/refractory B-cell cell cancers. This study will also look at whether 19(T2)28z1xx CAR T cells work against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Creatinine ≤2.0 mg/100 ml, direct bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x upper limit of normal (ULN)
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry.
* Histologically confirmed DLBCL and large B cell lymphoma, including

  * DLBCL, not otherwise specified (NOS), or
  * Transformed DLBCL from follicular lymphoma, or
  * High-grade B cell lymphoma (excluding Burkitt's lymphoma), or
  * Primary mediastinal large B cell lymphoma AND
  * Chemotherapy refractory disease, defined as a failure to achieve at least a partial response or disease progression within 12 months to the last therapy, OR
  * Disease progression or recurrence in ≤12 months of prior autologous stem cell transplant (ASCT), OR
  * Relapsed disease after 2 or more prior chemoimmunotherapies with at least one containing an anthracycline and CD20 directed therapy
* Patients need to have radiographically documented disease

Exclusion Criteria:

* ECOG performance status ≥2.
* Patients with active CNS disease
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Impaired cardiac function (LVEF <40%) as assessed by ECHO or MUGA scan.
* Patients with the following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction ≤6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration ≤6 months prior to enrollment
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible.
* Patients with prior allogeneic hematopoietic stem cell transplant are eligible, if more than 3 months from transplant and if patients have no active graft versus host disease (GvHD) and not on systemic immunosuppressive therapy.
* Prior CD19-directed therapy including CD19 CAR T cells is allowed, as long as expression of CD19 is confirmed by flow cytometry or immunohistochemistry.
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection are ineligible.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of the skin.
* Patients with presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, severe brain injuries are ineligible.
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) | 28 days post infusion
  Dose escalation will use a 3+3 design. DLT-evaluable participants are defined as those participants who were infused with 19(T2)28z1XX CAR T cells and who were monitored for toxicities during the first 28 days of post infusion.

SECONDARY OUTCOMES:
overall response rate (ORR) | 2 years
  Response and progression of the disease will be evaluated in this study using the Lugano Classification

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Park JH, Palomba ML, Perica K, Devlin SM, Shah G, Dahi PB, Lin RJ, Salles G, Scordo M, Nath K, Valtis YK, Lynch A, Cathcart E, Zhang H, Schoder H, Leithner D, Liotta K, Yu A, Stocker K, Li J, Dey A, Sellner L, Singh R, Sundaresan V, Tong X, Zhao F, Mansilla-Soto J, He C, Meyerson J, Hosszu K, McAvoy D, Wang X, Riviere I, Sadelain M. Results From First-in-Human Phase I Study of a Novel CD19-1XX Chimeric Antigen Receptor With Calibrated Signaling in Large B-Cell Lymphoma. J Clin Oncol. 2025 Jul 20;43(21):2418-2428. doi: 10.1200/JCO-24-02424. Epub 2025 Jan 30. PMID 39883889
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm